CLINICAL TRIAL: NCT05246995
Title: A Phase I, Open-label, Dose-escalation Study Evaluating the Safety, Tolerability, and Potential Efficacy of IBI325, an Anti-CD73 Antibody, Combined With Sintilimab in Patients With Advanced Solid Tumor
Brief Title: A Phase I Study of IBI325 in Patients With Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, Director of the hospital, Shandong Cancer Hospital and Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI325Y001
Record Dates: First submitted 2022-02-16; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI325 and Sintilimab combination does-escalation (Experimental)
  Interventions: Drug: IBI325+Sintilimab

INTERVENTIONS:
Drug: IBI325+Sintilimab — IBI325 + sintilimab combination does-escalation Patients will receive IBI325 monotherapy on Cycle 1 Day 1 ,and then receive IBI325 and sintilimab combination until progressive disease, intolerability, or other reasons leading to treatment discontinuation

SUMMARY:
The primary objective of this phase I study is to evaluate the safety and potential efficacy and to determine the recommended phase 2 dose (RP2D) of IBI325 combined with Sintilimab in patients with advanced solid tumors

ELIGIBILITY:
Inclusion

1. Histologically confirmed, locally advanced unresectable or metastatic tumors.
2. At least one measurable lesion per RECIST 1.1
3. Male or female subject at least 18 years old and no more than 75 years old.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) performance status 0 or 1.
5. Must have adequate organ function
6. Be able to provide archived or fresh tumor tissues Exclusion

1. Any anti-tumor treatment with 4 weeks, except anti-CD73 monoclonal antibody. 2. Subjects participating in another interventional clinical study, except for during the survival follow-up phase of the studies.

3. Unstable central nervous system netastases 4. Known active autoimmune disease or inflammatory disease 5. Known active infectious disease 6. Other uncontrolled systematic disease that may increase the risk of participating the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-23 (Estimated); Primary Completion 2023-03-23 (Estimated); Study Completion 2023-11-23 (Estimated)

PRIMARY OUTCOMES:
Number of patients with DLT | 42 days post first dose
  Number of patients who experienced a dose-limiting toxicity within the first 42 days after the first dose
Number of patients with treatment related AEs | Up to 90 days post last dose
  Number of patients who experienced a treatment related AEs from the first dose until 90days after the last dose

SECONDARY OUTCOMES:
Number of patients with response | Every 6 weeks until progressive disease or up to 24 months after treatment, whichever came first
  Number of patients with response per RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Province Cancer Hospital, Jinan, Shandong, China